CLINICAL TRIAL: NCT01101282
Title: Does the Addition of Positive Expiratory Pressure (PEP) Mask Therapy to Usual Medical Care Improve Patients' Symptoms, Quality or Life and Risk of Future Exacerbations in Individuals With Acute Exacerbations of Chronic Obstructive Pulmonary Disease (COPD)?
Brief Title: Does Positive Expiratory Pressure Mask Therapy Improve Recovery From Acute Exacerbations of Chronic Obstructive Pulmonary Disease?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: La Trobe University (Other)
Collaborators: The Alfred (Other); Austin Hospital, Melbourne Australia (Other)
Responsible Party: Principal Investigator, Christian Osadnik, Physiotherapist, PhD candidate, La Trobe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: (not yet specified)
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive
Keywords: PEP; exacerbation; physiotherapy; airway clearance; sputum; physical Therapy modalities
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 'Usual care' (No Intervention): Participants will receive 'usual medical care' consisting of the following:
  * Medical management: Bronchodilators, corticosteroids, antibiotics and supplemental oxygen will be provided (where appropriate) in accordance with Australian and New Zealand COPD management guidelines (COPDX guidelines).
  * Non-invasive ventilation: if clinically indicated and prescribed in accordance with standardised hospital guidelines.
  * Physical rehabilitation: Participants will be assessed by a physiotherapist and prescribed appropriate exercises to facilitate a safe and timely discharge. Participants will perform physical rehabilitation according to a standardised protocol with an aim of maximising physical function at discharge.
  * Other allied health (e.g. occupational therapy, speech pathology, dietician) assessments and interventions, as required.
- 'Usual care' plus PEP mask therapy (Experimental): This will comprise:
  * 'Usual care'
  * PEP mask therapy
  Interventions: Device: Positive expiratory pressure (PEP) mask therapy

INTERVENTIONS:
Device: Positive expiratory pressure (PEP) mask therapy — PEP mask therapy will be performed once/day, supervised, by an experienced physiotherapist until hospital discharge or ≥ 24 hours without sputum expectoration (whichever comes first). Written instructions shall also be provided, encouraging two more independent PEP mask sessions per day. Each session will comprise up to 5 cycles of 8-10 slightly active breaths, followed by 2 huffs (FET) and 2 coughs. A target pressure of 10-20 cms H20 during the middle of expiration shall be used (monitored via a pressure manometer).
  Arms: 'Usual care' plus PEP mask therapy

SUMMARY:
This study aims to identify whether the addition of positive expiratory pressure (PEP) mask therapy to standard medical care improves clinically important outcomes in individuals with acute exacerbations of chronic obstructive pulmonary disease. It is hypothesized that those who receive the additional PEP mask therapy will show greater improvements than those who do not.

DETAILED DESCRIPTION:
This study aims to identify whether the addition of positive expiratory pressure (PEP) mask therapy to standard medical care improves symptoms, quality of life and risk of re-exacerbation in individuals with acute exacerbations of chronic obstructive pulmonary disease.

A PEP mask is a small hand-held device that is self-applied over the nose and mouth. It creates a resistance against exhalation (outward) breaths which helps facilitate movement of sputum from the lungs towards the mouth.

Participants will be recruited from two tertiary metropolitan hospitals in Melbourne, Australia and randomised to receive either 'usual care' (comprising medical management, non-invasive ventilation if required, rehabilitation and allied health interventions) or 'usual care' plus PEP mask therapy for the duration of their hospital admission. All participants will then complete daily diaries for six months after discharge.

The effect of PEP mask therapy will be evaluated using a range of outcomes important to both patients and health care providers.

ELIGIBILITY:
Inclusion Criteria (all of the following criteria must be met):

* The primary reason for hospital admission is an acute exacerbation of clinically diagnosed COPD
* There is evidence of sputum expectoration or they are a chronic sputum producer ('regularly expectorates sputum on most days')
* They are able and willing to provide written, informed consent
* Recent (within the last 6 months) lung function data indicates obstructive lung disease (of any severity), according to the GOLD criteria: post-bronchodilator FEV1/FVC < 0.7 (only if available)
* They have a smoking history of ≥ 10 pack/years (only if diagnosis unclear)

Exclusion Criteria (none of the following criteria must be present):

* They are breathing via an artificial airway (e.g. endotracheal or tracheostomy tube)
* They have a more significant respiratory disease other than COPD (e.g. primary diagnosis of bronchiectasis, cystic fibrosis, interstitial lung disease, asthma, lung cancer)
* They have had recent (within the last 6 months) lung volume reduction procedure(s) (e.g. surgery, valve or stent insertion, or other), lung transplantation or pneumonectomy
* The intervention is contraindicated (including but not limited to evidence of undrained pneumothorax, significant frank haemoptysis, recent facial, oral, oesophageal or skull surgery/trauma, altered conscious state or inability to co-operate)
* They have poor oxygen saturation at rest (SpO2 < 88%) despite supplemental oxygen delivered via nasal prongs
* They intend to continue performing established ACT routines throughout the study period
* It is more than 48 hours since being admitted as an inpatient to hospital.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2010-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Symptom severity | Within 48 hours of presenting to hospital (day 1)
  Measured via the Breathlessness, Cough and Sputum Scale (BCSS).
Symptom severity | At hospital discharge (up to approx. day 10)
  Measured via the BCSS
Symptom severity | 8 weeks following hospital discharge
  Measured via the BCSS
Symptom severity | 6 months following hospital discharge
  Measured via the BCSS

SECONDARY OUTCOMES:
Disease-specific quality of life | Within 48 hours of presenting to hospital (day 1)
  Measured via the 4-week English (Australian) version of the St. George's Respiratory Questionnaire (SGRQ).
Disease-specific quality of life | 8 weeks following hospital discharge
  Measured via the SGRQ
Disease-specific quality of life | 6 months following hospital discharge
  Measured via the SGRQ
Need for assisted (non-invasive and/or invasive) ventilation during hospitalisation (within, and after 48 hours of presentation to hospital) | At hospital discharge (up to approx. day 10)
  The number of participants needing non-invasive or invasive ventilation during their inpatient stay shall be assessed. As early non-invasive ventilation is commonly used for the management of acute exacerbations of COPD, this outcome shall be assessed both within and after 48 hours of presentation to hospital. This aims to differentiate usual care from clinical deterioration.
Hospital length of stay | At hospital discharge (up to approx. day 10)
  Measured as number of days
Time to first exacerbation | 6 months following hospital discharge
  Measured as number of days
Time to first hospitalisation (due to respiratory illness) | 6 months following hospital discharge
  Measured as number of days
Number of acute exacerbations | 6 months following hospital discharge
  Measured as number of events
Number of hospitalisations (due to respiratory illness) | 6 months following hospital discharge
  Measured as number of events
Total number of hospitalised days | 6 months following hospital discharge
  Measured as number of hospitalised days
Lung function (spirometry) | At hospital discharge (up to approx. day 10)
  e.g. FEV1, FVC, FEV1/FVC%
Lung function (spirometry) | 6 months following hospital discharge
  e.g. FEV1, FVC, FEV1/FVC%
Mortality (actual, all cause) | At hospital discharge (up to approx. day 10)
  Measured as number of events
Mortality (actual, all cause) | 6 months following hospital discharge
  Measured as number of events
Mortality (predicted) | At hospital discharge (up to approx. day 10)
  Measured via calculation of the BODE index. The BODE index is derived from: Body mass index, Obstruction severity (spirometry), Dyspnoea (MRC dyspnoea scale) and Exercise tolerance (6 minute walk test).
Mortality (predicted) | 6 months following hospital discharge
  Measured via BODE index

CONTACTS AND LOCATIONS:
Overall Officials: Christian R Osadnik, Bachelor of Physiotherapy, Principal Investigator — La Trobe University
Locations (2):
- Australia (2):
  - The Austin Hospital, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria